CLINICAL TRIAL: NCT00586404
Title: Barrett's Esophagus Study (BEST) Trial - a Multi-Center and Endoscopic Outcomes Project
Brief Title: The Study of Barrett's Esophagus: What Are the Factors of Progression
Acronym: BEST
Status: Terminated | Type: Observational
Why Stopped: lack of enrollment
Sponsor: Midwest Biomedical Research Foundation (Other)
Collaborators: TAP Pharmaceutical Products Inc. (Industry); Kansas City Veteran Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, PRATEEK SHARMA, Principal Investigator, Midwest Biomedical Research Foundation
Organization: Midwest Veterans' Biomedical Research Foundation (Other)
Other Study IDs: PS0048
Record Dates: First submitted 2007-12-21; First posted 2008-01-04 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Barrett's Esophagus; Esophageal Neoplasms
Keywords: Barrett's Esophagus; Esophageal neoplasms; gastroesophageal reflux; gastrointestinal neoplasms
MeSH Terms: conditions — Barrett Esophagus; Esophageal Neoplasms; Gastroesophageal Reflux; Gastrointestinal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- A: Patients with confirmed Barrett's Esophagus

SUMMARY:
This trial is a multi-center clinical and endoscopic outcomes project involving a single large database of patients with Barrett's Esophagus (BE). The initial goal of this project is to define the incidence and prevalence of cancer and high-grade dysplasia (HGD) in patients with BE. Thus, our hypothesis is that systematic collection of data on the natural history of BE and risk factors for progression of BE will provide useful information to develop a decision model for risk stratification and risk reduction strategies in BE.

DETAILED DESCRIPTION:
Barrett's esophagus (BE) is defined as a change in the esophageal mucosa from normal squamous epithelium to columnar epithelium with intestinal metaplasia (1). There is compelling evidence that BE is a precursor lesion for adenocarcinoma of the esophagus (2). There is also evidence that the prevalence of BE is much higher than was initially suspected, and that the true incidence rate of cancer in patients with BE is much lower than previously estimated. Endoscopic surveillance of all patients with BE is not likely to be cost effective, or save many lives. Therefore, it is important to understand which patients with BE are likely to progress to malignancy, and equally important to determine which patients are not likely to progress.Because progression is an uncommon event, definitive studies of natural history including evaluation of numerous risk factors require large numbers of patients, that can only be accomplished in the context of a multicenter study. This model will be a useful tool leading to a reduction in overall health care costs.

An Opportunity to Generate the Essential Knowledge for Intervention. We have established an initial network of investigators interested in the 'Barrett's Esophagus Study' (a long term, longitudinal, prospective study) and collected preliminary data in patients with BE. To date, 1376 patients from 4 centers have been entered into a central databank. We have presented preliminary data on the incidence and prevalence rates of high-grade dysplasia and cancer at national meetings. We now propose the creation of a formal consortium to perform a cohort study with the ultimate primary aim of defining risk factors for the development of high-grade dysplasia and adenocarcinoma in patients with BE. Such a multi-center, prospective, cohort, multi-disciplinary approach to BE was endorsed by the "NIH PRG on stomach and esophageal cancers" (May 2002).

BACKGROUND & CLINICAL SIGNIFICANCE Barrett's Esophagus the pre-malignant lesion for esophageal adenocarcinoma - a Condition of Rapidly Increasing Incidence. Patients with BE are at an increased risk for the development of esophageal adenocarcinoma and esophagogastric junction adenocarcinoma. Adenocarcinoma of the esophagus is believed to arise from BE in a step-wise progression from low-grade dysplasia to high-grade dysplasia, finally leading to frank adenocarcinoma (4,5). The cost effectiveness of surveillance endoscopy in patients with BE is very sensitive to the incidence of cancer (11). The exact incidence of adenocarcinoma in patients with BE is not known and has been reported to vary from 1 in 50 patient-years of follow up to 1 in 285 patient-years of follow up (18-22). The published incidence data from existing cohorts of patients with BE have been influenced by the small number of patients being evaluated, short duration of follow-up as well as by the demographics of the population being studied (e.g. older patients, male sex). To date, the maximum number of patients included in a published study determining the incidence of adenocarcinoma has been only 327 patients (23,24). The ultimate goal of the proposed study is to establish a large cohort of patients with BE to address issues of incidence, progression and risk factors influencing progression. Such an approach was recently endorsed by the "NIH 2002 PRG on stomach and esophageal cancers".

Factors predicting the development of dysplasia and cancer in BE patients are unknown. A few possible factors have been associated with esophageal adenocarcinoma, but not studied in BE patients. These include GERD symptoms, obesity, diet, smoking, prior cholecystectomy, drugs and H pylori infection (negative association) (25-36). The presence of hiatal hernia and BE length have been associated with dysplasia and cancer development in BE patients in a preliminary single center study (37). Reflux symptoms have also been reported to be significantly more prevalent among parents and siblings of patients with BE and esophageal adenocarcinoma than spouse control relatives (38). A few uncontrolled reports have provided conflicting results on the role of anti-reflux surgery and the use of acid suppressive medications (proton pump inhibitors, H2 receptor antagonists) and their effect on the neoplastic progression in BE patients (39-43). However, all the studies to date in BE patients have been limited by small sample sizes, univariate analysis, short duration of follow-up, lack of adjustment for confounding variables etc. In this proposed study, risk factors and mechanisms of capturing data at each site and data transfer to the main study database will be discussed and implemented. Sample size calculations for appropriate univariate and multiple logistic regression analysis will be performed.

Proposed Study will Fill Significant Gaps in Knowledge. In the recent "NIH PRG on stomach and esophageal cancers (May 2002)" and a workshop sponsored by the NIH & The American Digestive Health Foundation on endoscopic priorities (44), experts in the field acknowledged that there was a need for multi-center, longitudinal, studies and there were significant gaps in the knowledge base of BE including:

1. Risk stratification of cancer risk
2. Appropriate method of surveillance and technique for identifying dysplasia
3. Frequency and benefits of surveillance
4. Optimal management of BE such as acid suppression and endoscopic reversal techniques The ultimate goal of the BE Study is to address issues #1 and #3 i.e. risk stratification of Barrett's patients, and by developing a large, multi-site database, will prepare the way for future studies that can address the other key issues.

The information gained will be clinically useful. We will define the natural history of progression of BE patients and to determine factors involved in this progression to high-grade dysplasia and cancer. The potentially unique answers obtained from the study would have major clinical relevance in

* Defining the natural history of dysplasia/cancer in BE patients and to identify risk factors involved in progression to dysplasia/cancer.
* Helping clarify what predisposes only a small subset of BE patients to develop dysplasia/cancer. Rigorous examination of a number of risk factors may define this patient group, thereby focusing our limited health care resources to the patient subset at increased risk for the development of dysplasia/cancer - "reduction in health care costs"
* Potential to change our current costly clinical practice of endoscopic surveillance of all BE patients, by limiting surveillance to the 'high-risk group' - "improve clinical decision making"
* Providing better and accurate information to our BE patients regarding their 'true' risk for dysplasia and cancer.

PRELIMINARY STUDIES At this time, preliminary data have been collected from the 4 participating centers, and merged into one single databank. These preliminary results were presented at the plenary sessions (45,46) of the American Gastroenterological Association (AGA) annual meeting in Atlanta, GA (May 2001) and at the American College of Gastroenterology (ACG) annual meeting in Las Vegas, NV (October 2001), indicating a common interest amongst the investigators and capability of working together.

Distribution of Degree of Dysplasia. From the four participating centers, 1376 patients have met the study criteria and had at least one endoscopy with biopsy revealing intestinal metaplasia, thus confirming the diagnosis of BE. At the initial endoscopy, the distribution of dysplasia was as follows:

Diagnosis Number of pts. Prevalence Low-grade dysplasia (LGD) 101 7.3% High-grade dysplasia (HGD) 42 3% Esophageal adenocarcinoma 91 6.7% Incidence and progression to low-grade dysplasia, high-grade dysplasia and esophageal adenocarcinoma. 1376 patients were enrolled in the prevalence phase of the study. To date, 618 patients (95% Caucasians, 14% Females) have had follow-up endoscopic procedures to examine the incidence of dysplasia/cancer. They have been followed for a total of 2546 patient-years; mean follow up 4.12 patient-years (range: 1-22.5 yrs). Twelve patients developed cancer during follow up for a cancer incidence of 1 in 212 patient-years of follow up or 0.5% per year. The mean time to development of cancer was 5.3 yrs (range: 2.4-11.2 yrs). Of interest, 7 of 12 patients had high-grade dysplasia before cancer development while 2 had only low-grade dysplasia; 3 developed cancer from BE without dysplasia documented at any point. 22 patients developed high-grade dysplasia during follow up for an estimate of high-grade dysplasia incidence of 1 in 116 patient-years of follow up or 0.9% per year. The mean time to high-grade dysplasia development was 3.8 yrs (range: 1.2-7.9 yrs). 11 of 22 patients developed high-grade dysplasia from BE without documented dysplasia, whereas the remaining 11 went from low-grade dysplasia to high-grade dysplasia.

Risk Factors for BE and adenocarcinoma. The epidemiology and natural history of BE has been poorly studied. Some factors have been associated with an increased risk for esophageal adenocarcinoma in the general population (see Table 1), but risk factors for progression in BE patients are not clear. A number of risk factors have been suggested as factors of risk in BE patients including age, gender, ethnicity, GERD symptoms, family history of BE/cancer, alcohol, tobacco, dietary factors (fat intake, cereal fiber, calcium etc.) acid suppressive medications, biomarkers, genetic markers etc. Given this long list of possible risk factors, we propose to convene a panel of experts in a planning committee to serve as jury in order to determine which of the potential risk factors should be measured in a prospective study and how they should be measured. This would narrow and refine the list of risk factors for the prospective study.

There are a lot of purported risk factors to be evaluated. Thus, there is a long list (see below) of potential factors of risk in patients with BE associated with progression to dysplasia and/or cancer:

(1) Age (2) Gender (3) Ethnicity (4) Reflux symptoms (5) Smoking (6) Alcohol (7) Dietary fat (8) Dietary fiber, vegetables, fruits (9) Dietary calcium (10) Obesity (11) Family history of reflux, BE or esophageal cancer (12) Use of aspirin, non-steroidal anti-inflammatory drugs (13) Use of lower esophageal sphincter relaxing medications (14) Use of acid suppressive medications (15) Cholecystectomy (16) Anti-reflux surgery (fundoplication) (17) Length of BE (18) Hiatal hernia (19) Helicobacter pylori infection (20) Low-grade dysplasia on biopsy This proposal will make it feasible to narrow on the factors to be studied in the prospective trial.

Statistical Analysis Prevalence and incidence rates: We expect to increase the baseline-screened population from 1376 to more than 2500 individuals in the final study. The number of patients we expect to enroll each year will be calculated and the expected number of new prevalence cases using the 9.7% prevalence rate with the preliminary study data will be estimated. In the preliminary study to date 618 patients have had at least one follow-up visit. Including the remaining 700 patients from the preliminary study and assuming a 10% rate for loss to follow up, we will have 6100-7450 patient years of follow up. The expected number of new incidence cases using the 1.3% incidence rate with the preliminary study data will be estimated.

ELIGIBILITY:
Inclusion Criteria:

* Sex: Male and female
* Age: 18-80 years
* Confirmed BE.

Exclusion Criteria:

* Columnar mucosa in the distal esophagus but no intestinal metaplasia on biopsy.
* Patients with BE who have undergone endoscopic ablation therapy or enrolled in chemoprevention trials. Since this is a natural history study, patients enrolled in intervention trials (e.g. those undergoing endoscopic ablation of their BE) will be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who have histologically confirmed Barrett's Esophagus
Sampling Method: Probability Sample
Enrollment: 1250 (Actual)
Dates: Start 2007-11 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
To determine the prevalence and incidence of low grade dysplasia, high grade dysplasia and adenocarcinoma in a large cohort of patients with Barrett's esophagus | up to 10 years

SECONDARY OUTCOMES:
To determine the magnitude of the contribution of selected factors (e.g. age, gender, ethnicity, obesity, tobacco use, alcohol use, ASA/NSAID/PPI use, duration of GERD symptoms, length of BE, HH) to the risk of HGD and CA | up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Prateek Sharma, MD, Principal Investigator — Department of Veterans Affairs Medical Center of Kansas City
Locations (4):
- United States (4):
  - Southern Arizona VA Medical Center, Tucson, Arizona
  - Bethesda Naval Medical Center, Bethesda, Maryland
  - Department of Veterans Affairs Medical Center, Kansas City, Missouri
  - Cleveland Clinic, Cleveland, Ohio

REFERENCES:
- [Background] Weinstein WM, Ippoliti AF. The diagnosis of Barrett's esophagus: goblets, goblets, goblets. Gastrointest Endosc. 1996 Jul;44(1):91-5. doi: 10.1016/s0016-5107(96)70239-0. No abstract available. PMID 8836727
- [Background] Shaheen NJ, Crosby MA, Bozymski EM, Sandler RS. Is there publication bias in the reporting of cancer risk in Barrett's esophagus? Gastroenterology. 2000 Aug;119(2):333-8. doi: 10.1053/gast.2000.9302. PMID 10930368
- [Background] Sampliner RE. Practice guidelines on the diagnosis, surveillance, and therapy of Barrett's esophagus. The Practice Parameters Committee of the American College of Gastroenterology. Am J Gastroenterol. 1998 Jul;93(7):1028-32. doi: 10.1111/j.1572-0241.1998.00362.x. No abstract available. PMID 9672324
- [Background] Reid BJ, Barrett MT, Galipeau PC, Sanchez CA, Neshat K, Cowan DS, Levine DS. Barrett's esophagus: ordering the events that lead to cancer. Eur J Cancer Prev. 1996 Dec;5 Suppl 2:57-65. doi: 10.1097/00008469-199612002-00009. No abstract available. PMID 9061296
- [Background] Reid BJ, Haggitt RC, Rubin CE, Roth G, Surawicz CM, Van Belle G, Lewin K, Weinstein WM, Antonioli DA, Goldman H, et al. Observer variation in the diagnosis of dysplasia in Barrett's esophagus. Hum Pathol. 1988 Feb;19(2):166-78. doi: 10.1016/s0046-8177(88)80344-7. PMID 3343032
- [Background] Devesa SS, Blot WJ, Fraumeni JF Jr. Changing patterns in the incidence of esophageal and gastric carcinoma in the United States. Cancer. 1998 Nov 15;83(10):2049-53. PMID 9827707
- [Background] Blot WJ, Devesa SS, Kneller RW, Fraumeni JF Jr. Rising incidence of adenocarcinoma of the esophagus and gastric cardia. JAMA. 1991 Mar 13;265(10):1287-9. PMID 1995976
- [Background] van Sandick JW, van Lanschot JJ, Kuiken BW, Tytgat GN, Offerhaus GJ, Obertop H. Impact of endoscopic biopsy surveillance of Barrett's oesophagus on pathological stage and clinical outcome of Barrett's carcinoma. Gut. 1998 Aug;43(2):216-22. doi: 10.1136/gut.43.2.216. PMID 10189847
- [Background] Streitz JM Jr, Andrews CW Jr, Ellis FH Jr. Endoscopic surveillance of Barrett's esophagus. Does it help? J Thorac Cardiovasc Surg. 1993 Mar;105(3):383-7; discussion 387-8. PMID 8445916
- [Background] Peters JH, Clark GW, Ireland AP, Chandrasoma P, Smyrk TC, DeMeester TR. Outcome of adenocarcinoma arising in Barrett's esophagus in endoscopically surveyed and nonsurveyed patients. J Thorac Cardiovasc Surg. 1994 Nov;108(5):813-21; discussion 821-2. PMID 7967662
- [Background] Provenzale D, Schmitt C, Wong JB. Barrett's esophagus: a new look at surveillance based on emerging estimates of cancer risk. Am J Gastroenterol. 1999 Aug;94(8):2043-53. doi: 10.1111/j.1572-0241.1999.01276.x. PMID 10445526
- [Background] Sharma P. Controversies in Barrett's esophagus: management of high grade dysplasia. Semin Gastrointest Dis. 2001 Jan;12(1):26-32. PMID 11215852
- [Background] Levine DS, Haggitt RC, Blount PL, Rabinovitch PS, Rusch VW, Reid BJ. An endoscopic biopsy protocol can differentiate high-grade dysplasia from early adenocarcinoma in Barrett's esophagus. Gastroenterology. 1993 Jul;105(1):40-50. doi: 10.1016/0016-5085(93)90008-z. PMID 8514061
- [Background] Falk GW, Rice TW, Goldblum JR, Richter JE. Jumbo biopsy forceps protocol still misses unsuspected cancer in Barrett's esophagus with high-grade dysplasia. Gastrointest Endosc. 1999 Feb;49(2):170-6. doi: 10.1016/s0016-5107(99)70482-7. PMID 9925694
- [Background] Reid BJ, Blount PL, Feng Z, Levine DS. Optimizing endoscopic biopsy detection of early cancers in Barrett's high-grade dysplasia. Am J Gastroenterol. 2000 Nov;95(11):3089-96. doi: 10.1111/j.1572-0241.2000.03182.x. PMID 11095322
- [Background] Weston AP, Sharma P, Topalovski M, Richards R, Cherian R, Dixon A. Long-term follow-up of Barrett's high-grade dysplasia. Am J Gastroenterol. 2000 Aug;95(8):1888-93. doi: 10.1111/j.1572-0241.2000.02234.x. PMID 10950031
- [Background] Schnell TG, Sontag SJ, Chejfec G, Aranha G, Metz A, O'Connell S, Seidel UJ, Sonnenberg A. Long-term nonsurgical management of Barrett's esophagus with high-grade dysplasia. Gastroenterology. 2001 Jun;120(7):1607-19. doi: 10.1053/gast.2001.25065. PMID 11375943
- [Background] Hameeteman W, Tytgat GN, Houthoff HJ, van den Tweel JG. Barrett's esophagus: development of dysplasia and adenocarcinoma. Gastroenterology. 1989 May;96(5 Pt 1):1249-56. doi: 10.1016/s0016-5085(89)80011-3. PMID 2703113
- [Background] Robertson CS, Mayberry JF, Nicholson DA, James PD, Atkinson M. Value of endoscopic surveillance in the detection of neoplastic change in Barrett's oesophagus. Br J Surg. 1988 Aug;75(8):760-3. doi: 10.1002/bjs.1800750813. PMID 3167523
- [Background] Miros M, Kerlin P, Walker N. Only patients with dysplasia progress to adenocarcinoma in Barrett's oesophagus. Gut. 1991 Dec;32(12):1441-6. doi: 10.1136/gut.32.12.1441. PMID 1773946
- [Background] Drewitz DJ, Sampliner RE, Garewal HS. The incidence of adenocarcinoma in Barrett's esophagus: a prospective study of 170 patients followed 4.8 years. Am J Gastroenterol. 1997 Feb;92(2):212-5. PMID 9040193
- [Background] O'Connor JB, Falk GW, Richter JE. The incidence of adenocarcinoma and dysplasia in Barrett's esophagus: report on the Cleveland Clinic Barrett's Esophagus Registry. Am J Gastroenterol. 1999 Aug;94(8):2037-42. doi: 10.1111/j.1572-0241.1999.01275.x. PMID 10445525
- [Background] Rudolph RE, Vaughan TL, Storer BE, Haggitt RC, Rabinovitch PS, Levine DS, Reid BJ. Effect of segment length on risk for neoplastic progression in patients with Barrett esophagus. Ann Intern Med. 2000 Apr 18;132(8):612-20. doi: 10.7326/0003-4819-132-8-200004180-00003. PMID 10766679
- [Background] Reid BJ, Levine DS, Longton G, Blount PL, Rabinovitch PS. Predictors of progression to cancer in Barrett's esophagus: baseline histology and flow cytometry identify low- and high-risk patient subsets. Am J Gastroenterol. 2000 Jul;95(7):1669-76. doi: 10.1111/j.1572-0241.2000.02196.x. PMID 10925966
- [Background] Funkhouser EM, Sharp GB. Aspirin and reduced risk of esophageal carcinoma. Cancer. 1995 Oct 1;76(7):1116-9. doi: 10.1002/1097-0142(19951001)76:73.0.co;2-i. PMID 8630885
- [Background] Farrow DC, Vaughan TL, Hansten PD, Stanford JL, Risch HA, Gammon MD, Chow WH, Dubrow R, Ahsan H, Mayne ST, Schoenberg JB, West AB, Rotterdam H, Fraumeni JF Jr, Blot WJ. Use of aspirin and other nonsteroidal anti-inflammatory drugs and risk of esophageal and gastric cancer. Cancer Epidemiol Biomarkers Prev. 1998 Feb;7(2):97-102. PMID 9488582
- [Background] Chow WH, Blot WJ, Vaughan TL, Risch HA, Gammon MD, Stanford JL, Dubrow R, Schoenberg JB, Mayne ST, Farrow DC, Ahsan H, West AB, Rotterdam H, Niwa S, Fraumeni JF Jr. Body mass index and risk of adenocarcinomas of the esophagus and gastric cardia. J Natl Cancer Inst. 1998 Jan 21;90(2):150-5. doi: 10.1093/jnci/90.2.150. PMID 9450576
- [Background] Lagergren J, Bergstrom R, Nyren O. Association between body mass and adenocarcinoma of the esophagus and gastric cardia. Ann Intern Med. 1999 Jun 1;130(11):883-90. doi: 10.7326/0003-4819-130-11-199906010-00003. PMID 10375336
- [Background] Gammon MD, Schoenberg JB, Ahsan H, Risch HA, Vaughan TL, Chow WH, Rotterdam H, West AB, Dubrow R, Stanford JL, Mayne ST, Farrow DC, Niwa S, Blot WJ, Fraumeni JF Jr. Tobacco, alcohol, and socioeconomic status and adenocarcinomas of the esophagus and gastric cardia. J Natl Cancer Inst. 1997 Sep 3;89(17):1277-84. doi: 10.1093/jnci/89.17.1277. PMID 9293918
- [Background] Chow WH, Blaser MJ, Blot WJ, Gammon MD, Vaughan TL, Risch HA, Perez-Perez GI, Schoenberg JB, Stanford JL, Rotterdam H, West AB, Fraumeni JF Jr. An inverse relation between cagA+ strains of Helicobacter pylori infection and risk of esophageal and gastric cardia adenocarcinoma. Cancer Res. 1998 Feb 15;58(4):588-90. PMID 9485003
- [Background] Vicari JJ, Peek RM, Falk GW, Goldblum JR, Easley KA, Schnell J, Perez-Perez GI, Halter SA, Rice TW, Blaser MJ, Richter JE. The seroprevalence of cagA-positive Helicobacter pylori strains in the spectrum of gastroesophageal reflux disease. Gastroenterology. 1998 Jul;115(1):50-7. doi: 10.1016/s0016-5085(98)70364-6. PMID 9649458
- [Background] Cameron AJ, Lomboy CT. Barrett's esophagus: age, prevalence, and extent of columnar epithelium. Gastroenterology. 1992 Oct;103(4):1241-5. doi: 10.1016/0016-5085(92)91510-b. PMID 1397881
- [Background] Gray MR, Donnelly RJ, Kingsnorth AN. The role of smoking and alcohol in metaplasia and cancer risk in Barrett's columnar lined oesophagus. Gut. 1993 Jun;34(6):727-31. doi: 10.1136/gut.34.6.727. PMID 8314502
- [Background] Lagergren J, Bergstrom R, Lindgren A, Nyren O. Symptomatic gastroesophageal reflux as a risk factor for esophageal adenocarcinoma. N Engl J Med. 1999 Mar 18;340(11):825-31. doi: 10.1056/NEJM199903183401101. PMID 10080844
- [Background] Lagergren J, Bergstrom R, Adami HO, Nyren O. Association between medications that relax the lower esophageal sphincter and risk for esophageal adenocarcinoma. Ann Intern Med. 2000 Aug 1;133(3):165-75. doi: 10.7326/0003-4819-133-3-200008010-00007. PMID 10906830
- [Background] Freedman J, Ye W, Naslund E, Lagergren J. Association between cholecystectomy and adenocarcinoma of the esophagus. Gastroenterology. 2001 Sep;121(3):548-53. doi: 10.1053/gast.2001.27217. PMID 11522738
- [Background] Weston AP, Badr AS, Hassanein RS. Prospective multivariate analysis of clinical, endoscopic, and histological factors predictive of the development of Barrett's multifocal high-grade dysplasia or adenocarcinoma. Am J Gastroenterol. 1999 Dec;94(12):3413-9. doi: 10.1111/j.1572-0241.1999.01602.x. PMID 10606296
- [Background] Romero Y, Cameron AJ, Locke GR 3rd, Schaid DJ, Slezak JM, Branch CD, Melton LJ 3rd. Familial aggregation of gastroesophageal reflux in patients with Barrett's esophagus and esophageal adenocarcinoma. Gastroenterology. 1997 Nov;113(5):1449-56. doi: 10.1053/gast.1997.v113.pm9352846.
- [Background] Katz D, Rothstein R, Schned A, Dunn J, Seaver K, Antonioli D. The development of dysplasia and adenocarcinoma during endoscopic surveillance of Barrett's esophagus. Am J Gastroenterol. 1998 Apr;93(4):536-41. doi: 10.1111/j.1572-0241.1998.161_b.x. PMID 9576444
- [Background] Sharma P, Sampliner RE, Camargo E. Normalization of esophageal pH with high-dose proton pump inhibitor therapy does not result in regression of Barrett's esophagus. Am J Gastroenterol. 1997 Apr;92(4):582-5. PMID 9128303
- [Background] McDonald ML, Trastek VF, Allen MS, Deschamps C, Pairolero PC, Pairolero PC. Barretts's esophagus: does an antireflux procedure reduce the need for endoscopic surveillance? J Thorac Cardiovasc Surg. 1996 Jun;111(6):1135-8; discussion 1139-40. doi: 10.1016/s0022-5223(96)70214-3. PMID 8642813
- [Background] Williamson WA, Ellis FH Jr, Gibb SP, Shahian DM, Aretz HT. Effect of antireflux operation on Barrett's mucosa. Ann Thorac Surg. 1990 Apr;49(4):537-41; discussion 541-2. doi: 10.1016/0003-4975(90)90298-k. PMID 2322047
- [Background] Csendes A, Braghetto I, Burdiles P, Puente G, Korn O, Diaz JC, Maluenda F. Long-term results of classic antireflux surgery in 152 patients with Barrett's esophagus: clinical, radiologic, endoscopic, manometric, and acid reflux test analysis before and late after operation. Surgery. 1998 Jun;123(6):645-57. PMID 9626315
- [Background] Lieberman D, Hamilton F. NIH-ADHF Workshop on Endoscopy Priorities: workshop statement and recommendations. American Digestive Health Foundation. Gastrointest Endosc. 1999 Mar;49(3 Pt 2):S3-4. doi: 10.1016/s0016-5107(99)70515-8. No abstract available. PMID 10049438
- [Background] 45. Sharma P, Reker D, Falk G, et al. Progression of Barrett's esophagus to high grade dysplasia and cancer - preliminary results of the Barrett's esophagus study trial. Gastroenterol 2001;120:A-16.
- [Background] 46. Sharma P, Weston AP, Falk G, Johnston M, Reker D, Sampliner RE. Can two upper endoscopies negative for dysplasia eliminate the need for future surveillance in patients with Barrett's esophagus? Am J Gastroenterol 2001;96:(Supplement)109.
- [Background] Cameron AJ, Zinsmeister AR, Ballard DJ, Carney JA. Prevalence of columnar-lined (Barrett's) esophagus. Comparison of population-based clinical and autopsy findings. Gastroenterology. 1990 Oct;99(4):918-22. doi: 10.1016/0016-5085(90)90607-3. PMID 2394347
- [Background] Kabat GC, Ng SK, Wynder EL. Tobacco, alcohol intake, and diet in relation to adenocarcinoma of the esophagus and gastric cardia. Cancer Causes Control. 1993 Mar;4(2):123-32. doi: 10.1007/BF00053153. PMID 8481491
- [Background] Brown LM, Swanson CA, Gridley G, Swanson GM, Schoenberg JB, Greenberg RS, Silverman DT, Pottern LM, Hayes RB, Schwartz AG, et al. Adenocarcinoma of the esophagus: role of obesity and diet. J Natl Cancer Inst. 1995 Jan 18;87(2):104-9. doi: 10.1093/jnci/87.2.104. PMID 7707381
- [Background] Kuczmarski RJ, Flegal KM, Campbell SM, Johnson CL. Increasing prevalence of overweight among US adults. The National Health and Nutrition Examination Surveys, 1960 to 1991. JAMA. 1994 Jul 20;272(3):205-11. doi: 10.1001/jama.272.3.205. PMID 8022039
- [Background] Terry P, Lagergren J, Hansen H, Wolk A, Nyren O. Fruit and vegetable consumption in the prevention of oesophageal and cardia cancers. Eur J Cancer Prev. 2001 Aug;10(4):365-9. doi: 10.1097/00008469-200108000-00010. PMID 11535879
- [Background] Terry P, Lagergren J, Ye W, Wolk A, Nyren O. Inverse association between intake of cereal fiber and risk of gastric cardia cancer. Gastroenterology. 2001 Feb;120(2):387-91. doi: 10.1053/gast.2001.21171. PMID 11159879
- [Background] Champion G, Richter JE, Vaezi MF, Singh S, Alexander R. Duodenogastroesophageal reflux: relationship to pH and importance in Barrett's esophagus. Gastroenterology. 1994 Sep;107(3):747-54. doi: 10.1016/0016-5085(94)90123-6. PMID 8076761
- [Background] Vaezi MF, Richter JE. Role of acid and duodenogastroesophageal reflux in gastroesophageal reflux disease. Gastroenterology. 1996 Nov;111(5):1192-9. doi: 10.1053/gast.1996.v111.pm8898632.
- [Background] Cameron AJ. Barrett's esophagus: prevalence and size of hiatal hernia. Am J Gastroenterol. 1999 Aug;94(8):2054-9. doi: 10.1111/j.1572-0241.1999.01277.x. PMID 10445527
- [Background] Montgomery E, Bronner MP, Goldblum JR, Greenson JK, Haber MM, Hart J, Lamps LW, Lauwers GY, Lazenby AJ, Lewin DN, Robert ME, Toledano AY, Shyr Y, Washington K. Reproducibility of the diagnosis of dysplasia in Barrett esophagus: a reaffirmation. Hum Pathol. 2001 Apr;32(4):368-78. doi: 10.1053/hupa.2001.23510. PMID 11331953
- [Background] 58. Rosner. Fundamental of Biostatistics, New York, NY: Duxberry Press 1995.
- [Background] 59. Hosmer, D.W. and S. Lemeshow. Applied Logistic Regression, New York, NY: John Wiley and Sons, 1989.
- [Background] 60. Allison, P. D. Logistic Regression using the SAS System, Theory and Applications. Cary, NC. SAS Institute Inc, 1999.
- [Background] 61. Harrell, F.E. Regression Modeling Strategies with Applications to Linear Models, Logistic Regression, and Survival Analysis. New York, NY Springer, 2001.
- [Background] Sharma P, Weston AP, Morales T, Topalovski M, Mayo MS, Sampliner RE. Relative risk of dysplasia for patients with intestinal metaplasia in the distal oesophagus and in the gastric cardia. Gut. 2000 Jan;46(1):9-13. doi: 10.1136/gut.46.1.9. PMID 10601047
- [Background] Weston AP, Krmpotich PT, Cherian R, Dixon A, Topalosvki M. Prospective long-term endoscopic and histological follow-up of short segment Barrett's esophagus: comparison with traditional long segment Barrett's esophagus. Am J Gastroenterol. 1997 Mar;92(3):407-13. PMID 9068459
- [Background] 64. Lipscomb SJ, Schoenfeld P, Johnston, Bethesda National Naval Med ctr, Bethesda. The incidence of high grade dysplasia and adenocarcinoma among patients with Barrett's esophagus: a cohort of 154 patients followed for a total of 471 patient-years. Gastroenterol 1999;116(4):A238.